CLINICAL TRIAL: NCT03726125
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic, and Glucodynamic Effects of LY3374849 in Healthy Subjects
Brief Title: A Study of LY3374849 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16939; I9R-MC-BSDA (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-10-03; First posted 2018-10-31 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10-15

CONDITIONS: Healthy
MeSH Terms: interventions — insulin degludec

STUDY DESIGN:
Intervention Model Description: Parts B and C are crossover design.
Who Masked: Participant, Investigator
Masking Description: Double-blind in Part A. Open label in Parts B and C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- LY3374849 - SC (Part A) (Experimental): Single subcutaneous (SC) dose of LY3374849
  Interventions: Drug: LY3374849 - SC
- Insulin Degludec - SC (Part A) (Experimental): Single SC dose of insulin degludec
  Interventions: Drug: Insulin Degludec - SC
- LY3374849 - SC (Part B) (Experimental): Single dose of LY3374849 administered SC in up to three of three study periods
  Interventions: Drug: LY3374849 - SC
- LY3374849 - IV (Part B) (Experimental): Single dose of LY3374849 administered intravenously (IV) in up to one of three study periods
  Interventions: Drug: LY3374849 - IV
- LY3374849 - IV (Part C) (Experimental): Single IV dose of LY3374849 in one of two study periods
  Interventions: Drug: LY3374849 - IV
- Insulin Degludec - IV (Part C) (Experimental): Single IV dose of insulin degludec in one of two study periods
  Interventions: Drug: Insulin Degludec - IV

INTERVENTIONS:
Drug: LY3374849 - SC — Administered SC
  Arms: LY3374849 - SC (Part A); LY3374849 - SC (Part B)
Drug: Insulin Degludec - SC — Administered SC
  Arms: Insulin Degludec - SC (Part A)
Drug: LY3374849 - IV — Administered IV
  Arms: LY3374849 - IV (Part B); LY3374849 - IV (Part C)
Drug: Insulin Degludec - IV — Administered IV
  Arms: Insulin Degludec - IV (Part C)

SUMMARY:
The aim of this trial is to evaluate the safety and tolerability of the study drug known as LY3374849, when given as an injection to healthy participants.

The study will also investigate how quickly the body absorbs and gets rid of LY3374849 and how it affects the levels of blood sugar in comparison to insulin degludec, after a single dose is given by injection under the skin and directly into a vein.

Participation in this study includes screening, which is required within 28 days before start of study and a follow up at least 28 days after receiving the last dose of study drug.

This study has 3 parts:

* Participants in Part A will complete 1 study period (approximately 1 week).
* Participants in Part B will complete 3 study periods (approximately 3 weeks).
* Participants in Part C will complete 2 study periods (approximately 2 weeks).

DETAILED DESCRIPTION:
Parts B and C added per protocol amendment, approved in April 2019.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or a female who cannot become pregnant
* Have a body mass index (BMI) of at least 18 kilogram per square meter (kg/m²)
* Have normal blood pressure, pulse rate, electrocardiogram (ECG), blood and urine laboratory test results that are acceptable for the study
* Have veins suitable for easy blood collection and glucose solution infusion

Exclusion Criteria:

* Are currently participating in or completed a clinical trial within the last 30 days or any other type of medical research judged to be incompatible with this study
* Had donated or had blood loss of more than 450 milliliters (mL) within the last 3 months
* Have a regular alcohol intake greater than 21 units/week (male), or 14 units/week (female)
* Smoke more than 10 cigarettes per day
* Are infected with hepatitis B or human immunodeficiency virus (HIV)
* Have a history of allergies or reactions to more than one drug, or significant severe drug allergy
* Are taking illegal drugs

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline up to study completion (estimated at 11 weeks)
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Glucodynamics: Total Amount of Glucose Infused (Gtot) | Baseline up to 36 hours post-dose for each study arm
  Glucodynamics: Gtot
Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3374849 | Baseline at predose through 6 days post-dose for each study arm
  Pharmacokinetics: AUC of LY3374849

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No